CLINICAL TRIAL: NCT01378637
Title: AMES Treatment of the Impaired Leg in Chronic Stroke Patients
Acronym: AMES
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AMES Technology (Industry)
Collaborators: Oregon Health and Science University (Other); Northwestern University (Other); Shirley Ryan AbilityLab (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7034; R44NS060192-03 (NIH)
Record Dates: First submitted 2011-02-18; First posted 2011-06-22 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Stroke; Cerebrovascular Accident; Hemiparesis
Keywords: Leg; Robotic device; AMES; Stroke; Cerebrovascular Accident; Rehabilitation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMES Leg treatment (Experimental): An investigational device flexes and extends the ankle over a range of 30 degrees while vibrators stimulate the tendons attached to muscles that move the foot. The subject's task is to assist the motion of the device by pulling or pushing with the foot. Feedback of ankle torque or the electrical signal produced by the muscles (EMG) while the subject is assisting the motion is provided during the 30 treatment sessions.
  Interventions: Device: AMES- Leg treatment

INTERVENTIONS:
Device: AMES- Leg treatment — 30 minutes of treatment of the leg consisting of the AMES device passively moving the ankle between plantarflexion and dorsiflexion with vibration of the tendons being stretched, while the participant tries to assist in the movement as much as possible.

SUMMARY:
The purpose of this protocol is to determine if individuals who had a stroke more than one year before entering the study and whose ankles remain substantially impaired are able to sense and move the affected leg better after 9-13 weeks of treatment with a robotic therapy device (AMES).

DETAILED DESCRIPTION:
Our research objective is to develop procedures to rehabilitate those stroke patients who, through conventional therapies, are not brought to a level of maximal recovery. The aims of the proposed project are to obtain a set of data from a total of 20 chronic stroke subjects, all with severe lower extremity disability, between the ages of 18-85, using a robotic therapeutic device placed in a rehabilitation clinic. This data will allow us to quantify the extent to which a combination of robotic-assisted exercise and tendon vibration from the AMES beta device induces secondary recovery from the effects of stroke on the lower extremity.

ELIGIBILITY:
Inclusion Criteria:

* Spastic hemiparesis
* At least 12 months post-stroke
* Can comfortably fit foot in treatment device
* Functioning proprioception
* Fugl-Meyer LE score >6 and <23
* Minimal hemi-neglect
* Observable volitional movement of the ankle in either plantar- or dorsi-flexion
* Cognitively and behaviorally capable of complying with the regimen

Exclusion Criteria:

* Fractures of treated limb resulting in loss of range of motion
* Spinal cord injury
* Deep venous thrombosis
* Peripheral nerve injury or neuropathy in the affected limb with motor disability
* Osteoarthritis limiting range of motion
* Uncontrolled high blood pressure/angina
* Exercise intolerant
* Skin condition not tolerant of device
* Progressive neurodegenerative disorder
* Uncontrolled seizure disorder
* Botox treatment within last 5 months
* Baclofen pump

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Motor Assessment of the Lower Affected Extremity | Measured three times: 1) Baseline; 2) After 30 Treatments (typically 10-13 weeks); and 3) Three Months after completing Treatments

SECONDARY OUTCOMES:
Gait Assessment | Measured three times: 1) Baseline; 2) After 30 Treatments (typically 10-13 weeks); and 3) Three Months after completing Treatments
  The gait assessment will consist of the timed 10-Meter walk and the Tinetti Gait Test.
Modified Ashworth Scale | Measured three times: 1) Baseline; 2) After 30 Treatments (typically 10-13 weeks); and 3) Three Months after completing Treatments
  Measurement of spasticity in the ankle joint.
Dynamic Balance/Weight Distribution | Measured three times: 1) Baseline; 2) After 30 Treatments (typically 10-13 weeks); and 3) Three Months after completing Treatments
  Measure the subject's right-left weight distribution and dynamic balance control.
Ankle Strength | Prior to each treatment session,
  Measurement of three attempts of dorsiflexion and three attempts of plantarflexion.
Passive Motion Test | Prior to each treatment session
  Measures the peak resistance in the affected ankle.
Active Range of Motion Test | Prior to each treatment session
  A joint tracking task guided by visual feedback on a computer screen.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Oken, MD, Principal Investigator — Oregon Health and Science University; Elliot Roth, MD, Principal Investigator — Northwestern University/Rehabilitation Institute of Chicago
Locations (2):
- United States (2):
  - Northwestern University/Rehabilitation Institute of Chicago, Chicago, Illinois
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No